CLINICAL TRIAL: NCT03377205
Title: Intramedullary Nailing Versus Plate Fixation of Ankle Fractures.
Brief Title: Intramedullary Nailing Versus Plate Fixation of Ankle Fractures. A Prospective, Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Ostfold Hospital Trust (Other); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Elisabeth Ellingsen Husebye, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/137 (REK)
Record Dates: First submitted 2017-03-21; First posted 2017-12-19 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plate (Active Comparator): Compression screws and neutralization plate.
  Interventions: Device: Compression screws and neutralization plate
- Intramedullary nail (Experimental): Acumed Fibular Rod System
  Interventions: Device: Acumed Fibular Rod System

INTERVENTIONS:
Device: Compression screws and neutralization plate — Open reduction and internal fixation with screws and plate
  Arms: Plate
Device: Acumed Fibular Rod System — intramedullary nailing of fibula
  Arms: Intramedullary nail

SUMMARY:
The purpose of this study is to make a survey of functional outcome, radiological outcome and complication rate after intramedullary nailing (IMN) and plate fixation of Weber B ankle fractures in elderly patients, and contribute in choosing the best surgical method for these ankle fractures.

DETAILED DESCRIPTION:
Open reduction and internal fixation (ORIF) is the gold standard treatment for unstable Weber B fractures, using compression screws and a neutralization plate. In the elderly, pre-existing co-morbidities, osteoporosis and poor skin conditions may give a high complication rate, including wound complications, symptomatic hardware and hardware failure. Due to concerns with complications related to ORIF, the technique with intramedullary fixation has been introduced. This method may simplify the management when poor skin conditions and osteoporotic bone, and has the potential to reduce the risk of soft tissue and hardware complications. Previous studies have showed that intramedullary fixation is probably the best choice for treating unstable ankle fractures in elderly patients, but more studies are needed to conclude the superiority to standard plate fixation.

ELIGIBILITY:
Inclusion Criteria:

* Acute unstable Weber B fracture (unimalleolar, bimalleolar or trimalleolar fractures).
* Operable with both methods of surgery within 3 weeks after injury.
* Men and women ≥ 60 yoa.

Exclusion Criteria:

* Prior injury or pathology with reduced ankle function.
* Other acute foot/ankle/leg injury that will affect ankle function.
* Fracture of the posterior malleolus that need fixation.
* Injury / pathology that may affect rehabilitation.
* Open fracture.
* Inoperable patient.
* Dementia (MMSE score ≤ 24 points), reduced competent to consent, not able to express himself/herself in Norwegian or English.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Society (AOFAS) score | 5 years
  Functional outcome as assessed by AOFAS score (0-100)

SECONDARY OUTCOMES:
Manchester-Oxford Foot questionnaire (MOxFQ) | 5 years
  Patient reported outcome as assessed by MOxFQ (0-100)
Olerud and Molander Score (OMS) | 5 years
  Patient reported outcome as assessed by OMS (0-100)
EuroQol-5d (Eq-5d) | 5 years
  Patient reported quality of life as assessed by Eq-5d index score
Visual analogue scale (VAS) | 5 years
  VAS scores for pain during rest (0-10), during walking (0-10), at night (0-10), and during daily activities (0-10), where 10 is best
Fracture reduction as assessed by CT scans | 3 months
  Number of patients with good, fair or poor fracture reduction
Malunion as assessed by CT scans | 5 years
  Number of patients with malunion
Nonunion as assessed by CT scans | 5 years
  Number of patients with nonunion
Osteoarthritis as assessed by CT scans | 5 years
  Number of patients with osteoarthritis assessed according to the criteria by McLennan et al
Infection | 3 months
  Number of patients with wound infection or deep infection
Delayed wound healing | 3 months
  Number of patients with delayed wound healing
Other complications | 5 years
  Number of patients with other complications (e.g. hardware complications, tromboemolism, neurologic complications, peroneus tendon irritation)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth E Husebye, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No